CLINICAL TRIAL: NCT01780012
Title: Secondary Prevention of Osteoporosis in Women Over 50 Years Old After Low Intensity Fracture of the Upper Limb: Evaluation of an Intervention Focused on the Patient.
Brief Title: Evaluation of an Osteoporosis Prevention Strategy in Women With Osteoporotic Fracture of the Upper Limb
Acronym: PREVOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PREVOST
Record Dates: First submitted 2013-01-28; First posted 2013-01-30 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis With Current Fragility Fracture
Keywords: osteoporosis; fragility fracture; secondary prevention
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Osteoporosis prevention program: Women will receive oral and written information and advices on osteoporosis, a letter and a leaflet on osteoporosis management to give to their family physician, and phone call reminders.
  Interventions: Behavioral: Osteoporosis prevention program
- Control (No Intervention): Control women will receive usual post-fracture care without information

INTERVENTIONS:
Behavioral: Osteoporosis prevention program — Women will receive an oral information and advices on osteoporosis, a written leaflet on osteoporosis (risk factors, diagnosis, prevention and treatments), a letter and a leaflet on osteoporosis management to give to their family physician and phone call reminders (D15, D30, D45) to advise them to consult their family physician and, if they have a BMD prescription, to perform their BMD
  Arms: Intervention

SUMMARY:
Osteoporosis is a disease characterized by reduced bone mass and increased skeletal fragility, predisposing to an increased fracture risk. The presence of a low trauma fracture is a powerful predictor of future fractures and about 50% of patients with a fragility fracture will suffer a subsequent fracture in the next 10 years (Center Jacqueline R, 2007). Osteoporotic fractures are associated with an increased morbidity and mortality but also high financial costs. However, less than 20% of patients presenting a low trauma fracture receive an appropriate post-fracture osteoporosis management (Little and Eccles, 2010). The hypothesis of a lack of information and an under assessment of consequences by both patients and physicians has been raised to explain this gap between recommended care and usual practices.

The aim of the PREVOST program is to assess the efficiency of patient-centered osteoporosis prevention program, after a fragility fracture of the upper limb, to improve post-fracture management of osteoporosis (ie BMD test and / or osteoporosis treatment) in women over 50 years old.

This open randomized controlled trial aims to compare the BMD or osteoporosis treatment prescription rate at 6 months after inclusion between two groups: "intervention" receiving information on fracture and osteoporosis (oral and written), phone call reminders and written information to give to their family physician, and "control" receiving usual care without information.

ELIGIBILITY:
Inclusion Criteria:

* Women aged over 50 years
* with a fragility fracture of wrist or humerus that occurred in the past 6 months
* treated in an emergency department or orthopedic department
* who signed the consent form

Exclusion Criteria:

* no signed consent
* previous history of femoral neck fracture
* poly-trauma or accident
* patients under osteoporosis treatment
* patients who performed a BMD test in the past 6 months
* patients with severe renal impairment, hyperthyroidism, bone primary or secondary malignancy.
* legal disability
* difficulty in understanding French
* psychiatric disorder

Ages: 50 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2012-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Proportion of women in the 2 groups who initiated a management of osteoporosis at 6 months (BMD or osteoporosis treatment prescription). | 6 months after inclusion
  At 6 months, women will be asked whether or not they received a BMD test prescription and/or an osteoporosis treatment prescription by their physician.

SECONDARY OUTCOMES:
Proportion of women in the two groups who performed BMD at 6 months | 6 months after inclusion
  At 6 months, women who received a BMD prescription will be asked whether or not they performed a BMD test; if they realized a BMD test, their result will be asked.
Proportion of women in the two groups with an increased perception of fracture risk. | 6 months after inclusion
  Women will answer the same questionnaire at inclusion and at 6 months to assess their fracture risk perception.
Proportion of women in the two groups who changed their behaviour in order to prevent future fractures: regular practice of physical activity, dairy products consumption and calcium and vitamin D supplementation. | 6 months after inclusion.
  Women will answer the same questionnaire at inclusion and at 6 months to assess their behaviour towards fracture risk or prevention of osteoporosis: physical activity, dairy products consumption and calcium and vitamin D supplementation
Proportion of women who improved their knowledge about osteoporosis | 6 months after inclusion
  Women will answer the same questionnaire at inclusion and at 6 months to assess their osteoporosis perception and knowledge (risk factors, severity,consequences, treatments)

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle IMER, Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Merle B, Chapurlat R, Vignot E, Thomas T, Haesebaert J, Schott AM. Post-fracture care: do we need to educate patients rather than doctors? The PREVOST randomized controlled trial. Osteoporos Int. 2017 May;28(5):1549-1558. doi: 10.1007/s00198-017-3953-z. Epub 2017 Feb 28. PMID 28246884